CLINICAL TRIAL: NCT04625231
Title: Shared Decision-Making Tool for Opioid Prescribing After Ambulatory Orthopedic Surgery in Veterans - A Randomized Controlled Clinical Trial
Brief Title: Shared Decision-Making Tool for Opioid Prescribing After Ambulatory Hand Surgery in Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-0160
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Opioid Use; Surgery
Keywords: orthopedics; hand surgery; opioid use; counseling; education

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both patients and investigators were blinded to group assignment until an envelope was opened after the patient consented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared-Decision Making Tool Group (Experimental)
  Interventions: Behavioral: Educational Shared-Decision Making Tool
- Standard of Care Group (No Intervention)

INTERVENTIONS:
Behavioral: Educational Shared-Decision Making Tool — Patients received a short video presentation on pain management, use of over the counter medication, side effects of opioids and over-the-counter medications and ability to choose the amount of opioid pills up to the standard care amount.
  Arms: Shared-Decision Making Tool Group

SUMMARY:
The purpose of this study is to determine if an educational patient-centered presentation reduced the amount of opioid pills requested and utilized by patients compared to standard of care group.

ELIGIBILITY:
* 1. Inclusion Criteria:
* a. 18-89 years of age
* b. Patient at the Orthopedic Department at the Veterans Health Administration
* c. Indicated for upper extremity surgeries: E.g., Carpal Tunnel Release, Trigger Finger Release, Cubital Tunnel Release, Ganglion Cyst Excision
* 2. Exclusion Criteria:
* a. History of opioid use disorder
* b. Had any recent surgery within four weeks of upper extremity procedure
* c. Taking opioids prior to surgery
* d. Returning to an institutionalized setting
* e. Pregnancy
* f. Unable to communicate in the English language
* g. Allergy to any medication recommended for post-operative analgesia

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Number of Opioid Pills Dispensed | 1 day (Once after surgery)
Number of Opioid Pills Consumed | 4 weeks

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System Pain Interference Score | Once a week for 4 weeks after surgery
  Lower scores are better
Patient-Reported Outcomes Measurement Information System Pain Intensity Score | Once a week for 4 weeks after surgery
  Lower scores are better

CONTACTS AND LOCATIONS:
Overall Officials: Rajshri Bolson, MD, Principal Investigator — Rocky Mountain Regional VA Medical Center
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No